CLINICAL TRIAL: NCT06300892
Title: Surgical Site Infections and the Microbiome: Understanding the Pathogenesis of Surgical Site Infections
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: SURG-2023-31841
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Open GI Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — samples from the incision site and GI tract
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing open GI surgery: Patients with SSI
  Interventions: Other: No intervention
- Control group: age-, sex-, diagnosis-, and wound class-matched control patients without SSI
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — samples from the incision site and GI tract collected

SUMMARY:
This is a prospective, observational study of patients undergoing open GI surgery. At the time of operation, samples will be collected from the incision site and GI tract. The study will follow patients up to 30 days postoperatively, monitoring for signs of SSI. Samples will be taken from all patients who develop SSI. Sequencing will be performed on a subset of samples based on our specific aims.

* Aim 1: conduct a case-control study of patients with SSI and age-, sex-, diagnosis-, and wound class-matched control patients without SSI, comparing microbiome alpha diversity and community composition with 16S RNA sequencing to determine the association with SSI.
* Aim 2: identify the strain of bacteria isolated from SSIs using shotgun metagenomic sequencing and determine whether the specific strain was present in the skin and gut at the time of operation.

ELIGIBILITY:
Inclusion Criteria:

* We will include adult patients (age ≥ 18 years)
* Undergoing open abdominal surgery during the study period.
* Open abdominal surgery will include any abdominal procedure entering the peritoneal cavity through a midline incision with a skin incision that is 5cm or greater.

Exclusion Criteria:

* Patients with planned minimally invasive surgery including laparoscopic or robotic surgery as these patients have lower rates of surgical site infections (SSIs). Patients who have a laparoscopic or robotic surgery converted to open surgery will be excluded.
* Appendectomy and cholecystectomy as these patients have lower risk of SSI.
* Vascular, gynecological, obstetric, urological or transplantation.
* Trauma patients.
* Patients without source control at the index operation including those with an open abdomen, no fascial closure, or temporary abdominal closure device (such as abthera dressing).
* Pediatric patients (age<18 years).
* Patients who decline swab/specimen collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults over the age of 18 years, who are undergoing open abdominal surgery with a midline incision.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
alpha diversity composition | Baseline, Day 30 post-op
  Alpha diversity composition at the surgical incision site at multiple time points
microbial community composition | Baseline, Day 30 post-op
  microbial community composition at the surgical incision site at multiple time points
pathogenic strain of bacteria | Baseline, Day 30 post-op
  Pathogenic strain of bacteria at SSI compared with pathogens isolated from skin and/or GI tract microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Rickard, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States